CLINICAL TRIAL: NCT02638649
Title: Prehospital Use of Ultrasound in Undifferentiated Shortness of Breath
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1511016808
Record Dates: First submitted 2015-12-11; First posted 2015-12-23 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pneumonia; Pulmonary Edema; Dyspnea
Keywords: lung ultrasound
MeSH Terms: conditions — Pneumonia; Pulmonary Edema; Dyspnea | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- subjects who call 911 for dyspnea: All subjects who call 9-1-1 for difficulty breathing will have the potential to be enrolled in the study.
  Interventions: Procedure: Lung ultrasound; Device: ultrasound

INTERVENTIONS:
Procedure: Lung ultrasound — At each call, the paramedic will initially evaluate the patient clinically conducting a standard history and physical exam. The paramedic will then use the portable U/S machine to look for the presence of either unilateral or bilateral B-lines indicating possible pneumonia (in the case of unilateral B-lines) or pulmonary edema (in the case of bilateral B-lines). The paramedic will then document the presence or absence of B-lines for each lung on the prehospital study sheet. The paramedic will then use the U/S to evaluate for the presence of pleural effusions, lung sliding and pericardial effusion.
Device: ultrasound

SUMMARY:
This is a pilot observational feasibility study of the ability of paramedics to assess thoracic ultrasound findings in the prehospital environment. The primary goal of the study is to determine whether paramedics are able to accurately assess for sonographic B-lines in patients with undifferentiated shortness of breath at least 80% of the time in the prehospital environment using a portable ultrasound (U/S) device.

DETAILED DESCRIPTION:
In the first phase of the study, a cohort of senior and supervisory paramedics will be recruited into the study. These paramedics would undergo didactic and hands-on training to learn how to operate the U/S machine, and obtain and interpret basic U/S images. The paramedics will then participate in video review sessions and spend time in the emergency department (ED) with the U/S team to get hands-on experience with patients. In the second phase of the study, paramedics will be staffing ambulances or fly cars in and around the greater New Haven region and will respond to dyspnea calls. At each call, the paramedic will initially evaluate the patient clinically conducting a standard history and physical exam. The paramedic will then use the portable U/S machine to look for the presence of either unilateral or bilateral B-lines indicating possible pneumonia (in the case of unilateral B-lines) or pulmonary edema (in the case of bilateral B-lines). The paramedic will then document the presence or absence of B-lines for each lung on the prehospital study sheet. The paramedic will then use the U/S to evaluate for the presence of pleural effusions, lung sliding and pericardial effusion.

ELIGIBILITY:
Inclusion Criteria:

- Dyspnea and any of the following:

* Respiratory rate > 20
* Room air oxygen saturation < 92%
* Accessory muscle use, tripod position, nasal flaring
* Exam with evidence of rales/rhonchi or wheezing
* In acute respiratory distress on paramedic evaluation
* Any patient in acute respiratory distress with

Exclusion Criteria:

* Trauma
* Burns
* Pregnancy
* Kussmaul respirations from metabolic acidosis
* Cheyne-stokes from increased ICP (intracranial pressure), heart failure or CVA
* Drowning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of Paramedics' assessments of ultrasound for unilateral or bilateral B-lines | up to 12 months
  The paramedic will use the portable U/S machine to look for the presence of either unilateral/bilateral B-lines indicating possible pneumonia (unilateral B-lines) or pulmonary edema (bilateral B-lines). The paramedic will document the presence or absence of B-lines for each lung on the prehospital study sheet. The attending ED physician will be notified of the enrolled patient and, blinded to the paramedic's interpretation, will then conduct the same U/S study and document their findings and the final diagnosis of the patient using the patient's name, birthdate and MRN (Medical Record Number) on the ED study sheet. An U/S expert, blinded to the patient's diagnosis, the U/S operator, and confirmatory imaging, will review the recorded images obtained in the prehospital setting. The expert's interpretation of the images will be confirmed by a second expert for at least 15 % of the cases. The goal is 80% accuracy. The accuracy will be evaluated up to 12 months after the U/S is taken.

SECONDARY OUTCOMES:
Accuracy of Paramedics' assessments of ultrasound for interpretation of lung sliding, pleural effusions, and pericardial effusions. | up to 12 months
  The paramedic will use the U/S to evaluate for the presence of pleural effusions, lung sliding and pericardial effusion. The attending ED physician will be notified of the enrolled patient and, without knowing the paramedic's interpretation, will then conduct the same U/S study and document his or her findings and the final diagnosis of the patient using the patient's name, birthdate and MRN on the ED study sheet. An U/S expert, blinded to the patient's diagnosis, the U/S operator, and confirmatory imaging, will review the recorded images obtained in the prehospital setting. The expert's interpretation of the images will be confirmed by a second expert for at least 15 % of the cases. The goal is 80% accuracy. The accuracy will be evaluated up to 12 months after the ultrasound has been taken.

CONTACTS AND LOCATIONS:
Overall Officials: David C Cone, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale-New Haven Hospital-Saint Raphael Campus, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No